CLINICAL TRIAL: NCT05122247
Title: Generalizable Machine Learning to Predict Acute Care During Outpatient Systemic Cancer
Brief Title: Machine Learning to Predict Acute Care During Cancer Therapy
Acronym: Chemo-SHIELD
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00109633
Record Dates: First submitted 2021-11-05; First posted 2021-11-16 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Chemotherapeutic Toxicity
Keywords: machine learning; algorithm; outpatient
MeSH Terms: interventions — Machine Learning Algorithms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Machine learning algorithm — machine learning directed identification of chemotherapy patients at high-risk for emergency department acute care and/or hospitalization

SUMMARY:
The objective of this study is to apply a validated machine-learning based model (SHIELD-RT, NCT04277650) to a cohort of patients undergoing systemic therapy as outpatient cancer treatment to generate an automatic system for the prediction of unplanned hospital admission rates and emergency department encounters.

DETAILED DESCRIPTION:
A previously described machine learning (ML)-based model accurately predicted ED visits or hospitalizations for cancer patients undergoing radiation therapy or chemoradiation. An IRB approved prospective randomized trial, SHIELD-RT (NCT04277650) found that preemptive intervention for patients undergoing radiation and chemoradiation based on the ML model's risk stratification decreased the relative risk of acute care visits by 50%, showing that ML-guided escalation of care improved personalized supportive care and treatment compliance while decreasing healthcare costs.

The objective of this study is to apply this validated ML based model to a cohort of patients undergoing systemic therapy as outpatient cancer treatment to generate an automatic system for the prediction of unplanned hospital admission rates and emergency department encounters. Once validated, this study will add to the previously published body of evidence supporting a randomized trial evaluating the ML algorithm's ability to assign intervention for patients receiving systemic therapy at highest risk for acute care encounters.

ELIGIBILITY:
Inclusion Criteria:

* had treatment encounter in the Duke Medical Oncology department from January 7th, 2019 to June 30th, 2019
* DUHS medical record available

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Duke patients undergoing chemotherapy who had at least one treatment encounter between 1/7/2019 and 6/30/2019
Sampling Method: Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
number of unplanned of hospital admission or emergency department visits during systemic therapy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Palta, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hong JC, Eclov NCW, Dalal NH, Thomas SM, Stephens SJ, Malicki M, Shields S, Cobb A, Mowery YM, Niedzwiecki D, Tenenbaum JD, Palta M. System for High-Intensity Evaluation During Radiation Therapy (SHIELD-RT): A Prospective Randomized Study of Machine Learning-Directed Clinical Evaluations During Radiation and Chemoradiation. J Clin Oncol. 2020 Nov 1;38(31):3652-3661. doi: 10.1200/JCO.20.01688. Epub 2020 Sep 4. PMID 32886536